CLINICAL TRIAL: NCT06702826
Title: Efficacy and Safety of Cadonilimab Combined With Stereotactic Radiotherapy as Second-line Treatment for Brain Metastases From Non-small Cell Lung Cancer (NSCLC) : a Single-arm, Open-label, Phase II Clinical Trial
Brief Title: Cadonilimab Combined With Stereotactic Radiotherapy as Second-line Treatment for Brain Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rongrong Zhou (Other)
Responsible Party: Sponsor-Investigator, Rongrong Zhou, Deputy Director of Department of Oncology, Xiangya Hospital of Central South University
Organization: Xiangya Hospital of Central South University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202410188
Record Dates: First submitted 2024-11-18; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Non Small Cell Lung Cancer; Brain Metastases; Stereotactic Radiation; Immunotherapy
Keywords: non small cell lung cancer; brain metastases; SRS; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Spermine Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab combined with SRS (Experimental): Eligible subjects were treated with stereotactic radiotherapy for brain metastases plus Cadonilimab followed by maintenance therapy with Cadonilimab alone
  Interventions: Drug: Cadonilimab combined with SRS

INTERVENTIONS:
Drug: Cadonilimab combined with SRS — Eligible subjects were treated with stereotactic radiotherapy for brain metastases plus Cadonilimab followed by maintenance therapy with Cadonilimab alone

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of Cadonilimab combined with stereotactic radiation therapy in the second-line treatment of brain metastases from non-small cell lung cancer (NSCLC).

The main questions it aims to answer are:

* Does Cadonilimab combined with SRT in the second-line treatment of brain metastases provide better results?
* Is the toxicity of Cadonilimab combined with SRT manageable in second-line treatment of brain metastases? Researchers will compare evaluate the efficacy and safety of Cadonilimab combined with SRT as a second-line treatment for patients with advanced NSCLC：
* Receive Cadonilimab combined with SRT for brain lesions.
* Visit the hospital regularly once every 12 weeks for checkups and tests

DETAILED DESCRIPTION:
Lung cancer is the cancer with the highest morbidity and mortality in the world. The most common metastatic site of lung cancer is the brain.

Radiotherapy is a classic treatment for brain metastases from lung cancer. Stereotactic radiosurgery (SRS) has image-guided technology, which can accurately find the location of the tumor with an accuracy of millimeters, and effectively reduce the radiation to the surrounding normal tissues. According to the relevant recommendations of the NCCN guidelines for Central nervous System Tumors (first edition 2022), SRS can be given priority to patients with newly diagnosed localized brain metastases or with stable systemic tumor control, which can better protect the cognitive function of patients. SRS should be considered initial therapy in patients with a limited number of brain metastases. Citation (S) : SRS should be considered especially in patients with good physical activity status (PS) and small total tumor volume.

The brain was once considered to be an immune privilege organ, which can actively inhibit any immune response. The 2019 NCCN guidelines have recommended immune checkpoint inhibitors (ICIs) as the first-line treatment for some patients with lung cancer, and the application of ICIs in lung cancer with brain metastases is also being explored. Several phase III RCT studies have shown that immunotherapy prolongs the survival of patients with brain metastases.

As a classic treatment for brain metastases from lung cancer, radiotherapy can promote the anti-tumor immune effect by inducing immunogenic cell death, exposing tumor-associated antigens, activating dendritic cells, changing the tumor microenvironment, and enhancing the expression of intercellular adhesion molecule-1 (ICAM-1), Fas and major histocompatibility complex Ⅰ (MHCⅠ) in tumor cells. High-dose fractionated radiotherapy also has immunogenicity, which may open the blood-brain barrier (BBB) and promote the entry of ICI into brain tissue. However, radiotherapy can up-regulate the expression of PD-L1 and inhibit tumor immunity, which can be improved by ICI. In conclusion, intracranial radiotherapy combined with ICIs has feasibility and theoretical basis for the treatment of malignant tumors.

Cadonilimab is a bispecific antibody (BsAb) that can bind to both PD-1 and CTLA-4 with high affinity. It is a novel tumor immunotherapy drug with a quadrivalent structure and a short half-life, and has been shown to have less toxicity than the combination of anti-PD-1 and anti-CTLA-4 antibodies in monkey toxicity studies. These features make it possible that the use of Cadonilimab in cancer subjects may have better efficacy and safety.

In conclusion, the combination of Cadonilimab with radiotherapy has potential advantages and is expected to have the potential to further improve antitumor efficacy. Therefore, the aim of this study is to evaluate the efficacy and safety of Cadonilimab combined with SRS in the treatment of brain metastases from NSCLC, and to provide evidence for future studies.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ 75 years old; Both male and female;
2. ECOG 0-1;
3. Histologically or cytologically confirmed non-small cell lung cancer;
4. Progression with brain metastasis after previous first-line anti-tumor therapy;
5. Requirements for brain metastases: ① measurable brain metastases without radiotherapy; ②SRS/FSRT: the maximum tumor volume of brain metastases was less than 10cm3, the single diameter was less than 3cm, and the total volume of brain metastases involved was less than 15 cm3.
6. Response to previous checkpoint inhibitor therapy on the initial response assessment;
7. If a metastatic lesion of the head has been irradiated, the cumulative radiation dose does not exceed the tolerated dose to all structures.
8. For patients with measurable CNS lesions, the longest diameter on MRI images is ≥10mm, which is suitable for repeated and accurate measurement.
9. Subjects were evaluated for all extracranial disease sites (e.g., by computed tomography (CT) scan and bone scan or positron emission tomography (PET-CT) within 14 days before the first dose.
10. Subjects had to have a baseline brain MRI scan within 14 days before the first dose of medication.
11. Estimated survival time > 12 weeks.
12. Participants of childbearing age must agree to use effective contraception during the trial; In women of childbearing age, a serum or urine pregnancy test must be negative.
13. Patients who are not lactating.
14. Have definite and good organ functions:
15. Provide informed consent voluntarily, and be willing and able to comply with the follow-up, treatment, laboratory testing, and other study requirements specified in the study schedule.

Exclusion Criteria:

Subjects who meet any of the following criteria are not eligible to participate in the study:

1. Experienced grade 3-4 intracranial toxicity (pituitary or central nervous system toxicity);
2. No measurable intracranial metastatic lesions without radiotherapy;
3. Meningeal metastasis;
4. If receiving chemotherapy or targeted therapy, the washout period should not exceed 3 weeks; if receiving brain metastasis resection, the washout period should not exceed 2 weeks;
5. Have significant autoimmune diseases
6. Prior treatment with a cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) inhibitor.
7. Previous (within 5 years) or concurrent other malignant tumors
8. History of anaphylaxis to any monoclonal antibody and/or study drug component.
9. A history of or current noninfectious pneumonia/interstitial lung disease requiring systemic glucocorticoids.
10. Serious infection within 4 weeks before the first dose.
11. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
12. Subjects required systemic treatment with corticosteroids (>10mg prednisone equivalent per day) or other immunosuppressive drugs within 14 days before taking the study drug.
13. Patients with clinically significant cardiovascular disease
14. Enroll in another clinical study at the same time, unless it is an observational, noninterventional clinical study or a follow-up of an interventional study.
15. Received live vaccine within 30 days before the first dose, or planned to receive live vaccine during the study.
16. Known history of mental illness, substance abuse, alcohol or drug abuse.
17. Pregnant or lactating women.
18. The presence of any past or current medical conditions, treatments, or laboratory abnormalities may confound the results of the study, interfere with the full participation of the subject in the study, or may not be in the best interest of the subject to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
iORR | From date of enrollment until the date of first documented intracranial progression, assessed up to 2 years.
  Intracranial objective response rate (iORR) was defined as the proportion of patients who achieved a prespecified reduction in tumor volume and maintained the minimum time requirement, including CR and PR cases.

SECONDARY OUTCOMES:
PFS | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  Progression-free survival (PFS) : defined as the time from first use of a study drug to documentation of disease progression (according to RECIST v1.1) or death from any cause, whichever occurred first.
iPFS | From date of enrollment until the date of first documented intracranial progression or date of death from any cause, whichever came first, assessed up to 2 years
  Intracranial Progress Free Survival rate (iPFS) : the time from clinical detection of brain metastases to the first occurrence of intracranial progression or death. iPFS was assessed according to the Response Assessment of Brain Metastases in Neurooncology (RANO-BM) criteria.
OS | From date of enrollment until the date of death from any cause, whichever came first, assessed up to 2 years
  Overall survival (OS) : defined as time from treatment initiation to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China